CLINICAL TRIAL: NCT06257914
Title: ASICS: Aberrometry and Straylight Measurements as an Indication for Cataract Surgery
Brief Title: Aberrometry and Straylight Measurements as an Indication for Cataract Surgery
Acronym: ASICS
Status: Enrolling by invitation | Type: Observational
Sponsor: Amphia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N2024-0666
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-02

CONDITIONS: Cataracts; Cataract Surgery
Keywords: aberrometry; straylight; PROM; cataract; indication for cataract surgery
MeSH Terms: conditions — Cataract | interventions — Aberrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cataract: Patients with cataract in both eyes
  Interventions: Diagnostic Test: Catquest-9SF

INTERVENTIONS:
Diagnostic Test: Catquest-9SF — Measurement of self-assessed visual function with Catquest-9SF, measurement of ocular aberrations with iTrace (Tracey Technologies), and straylight measurements with C-Quant (Oculus)
  Other Names: Aberrometry (iTrace); Straylight measurement (C-Quant)

SUMMARY:
Cataracts are a clouding of the lens of the eye. Cataract surgery replaces the cloudy lens with a clear artificial lens. It is one of the leading causes of low vision worldwide. Since cataracts are mostly age-related, the number of patients with cataracts is increasing sharply due to an ageing population. The indication for cataract surgery is currently based on the visual impairment experienced by the patient, a measurement of visual acuity and the ophthalmologist's assessment of the extent to which the clouding of the lens explains the patient's symptoms.

It has been said that after cataract surgery, "the world opens up to you". However, about 10% of patients actually experience worse vision after surgery. This amounts to almost a whole month of potentially unnecessary surgery. It is therefore important to develop a more objective indicator for cataract surgery.

Our study focuses on measuring the optical quality of the eye before and after cataract surgery. The investigators also ask patients before and after cataract surgery how patients themselves perceive the quality of their vision. The investigators do this with different patient-reported outcomes. The investigators investigate whether the objective measurement of the optical quality of the eye can predict which patients will be satisfied with the cataract surgery. With this, the investigators aim to further improve patient care and prevent unnecessary surgery.

DETAILED DESCRIPTION:
Cataracts are a clouding of the lens of the eye. The symptoms of cataracts depend on where the clouding is in the lens and how extensive it is. Symptoms that patients may experience are blurred vision, poor vision at night, double vision in one eye, glare from backlight (such as from car headlights or a low sun), dulling of colours and a rapid change in refractive error. It is the most common cause of low vision in the world. Treatment for cataracts is surgical replacement of the cloudy lens for a clear artificial lens. The indication for cataract surgery is currently based on the visual impairment experienced by the patient, a measurement of visual acuity and the ophthalmologist's assessment of the extent to which the cloudiness of the lens explains the patient's symptoms.

Despite considering all these factors, it can be difficult for ophthalmologists to determine in advance which patient will benefit from cataract surgery. For example, visual acuity before surgery has been shown to be a poor indicator of cataract surgery outcome. There is also a limited relationship between the severity of clouding in the lens and the outcome of surgery. Questionnaires that assess patient-reported quality of vision (Patient Reported Outcome Measures, PROMs), such as the Catquest-9SF, also have limited predictability with regard to cataract surgery outcome. For example, the quality of vision of a significant number of patients who reported normal visual functioning before cataract surgery improves with surgery anyway.

In contrast, about 10% of all patients report that their visual functioning actually deteriorates with cataract surgery. There is also a limited correlation between how patients rate their change in visual functioning due to surgery in general (i.e., as much better, slightly better, no difference, slightly worse and much worse) and how patients report their visual functioning according to the Catquest-9SF. In other words, patients who report that their visual functioning after surgery felt much better than before sometimes report a worsening of their functioning with the Catquest-9SF questionnaire. It should be noted that the Catquest-9SF PROM is considered both clinically and scientifically the best questionnaire to measure change in visual functioning due to cataract surgery.

There are several reasons why patients may be dissatisfied after cataract surgery. In general, the more severe the discomfort caused by cataracts before surgery, the more satisfied patients are with the result obtained from the surgery. However, even a high percentage of patients with relatively few symptoms before surgery report having gained from the surgery after surgery. On the other hand, there is also a significant percentage of patients who deteriorate in visual function despite many complaints before surgery. The most commonly reported causes of dissatisfaction after cataract surgery with implantation of a standard artificial lens are dry eye and floaters. No research has been done on the extent to which these issues can be identified in advance.

Making the right indication for cataract surgery is important because surgery is irreversible. If the patient is dissatisfied with the result obtained, the old situation cannot be restored. Although the percentage of patients who are not satisfied after cataract surgery is small (10%), it is substantial in absolute numbers. The number of patients that is dissatisfied with the outcome of their cataract surgery corresponds to almost an entire month of cataract operations that, in retrospect, might better not have been performed.

A more objective and perhaps better indicator is based on the optical quality of the eye. Indeed, in essence, cataracts reduce the visual performance of the eye by deteriorating the optical quality of the lens. The optical quality of the eye is determined by optical aberrations and light scattering. Optical aberrations are deviations in the path that light rays travel that cause the light rays not to focus on a single point. These aberrations can be measured with an aberrometer. Light scattering is caused by small local irregularities in the refractive index in the ocular media. The visual effect of light scattering in the eye is straylight. This creates a veil of light over the retina, which reduces the contrast of the image projected on the retina. It also leads to glare from light. This can be measured with the C-Quant scattered light meter (www.oculus.de).

Aberrations and straylight complement each other. The optical quality of the eye is often expressed as the point spread function (PSF; in English, Point Spread Function). This function represents how a (point) light source is spread when it passes through the eye onto the retina. The central part of the PSF relates to optical aberrations; the peripheral part to light scattering. Vision is determined by the centre of the PSF.

Aberrometry and straylight measurements have been used independently to evaluate cataracts. Indeed, in cataracts, both the amount of aberrations and straylight increase. And both improve with cataract surgery. However, they have never been used together to predict the outcome of surgery. The closest is a study in which visual acuity and stray light were used as indicators of cataract surgery. In this study, the investigators showed that visual acuity and straylight contributed similarly to the predictive outcome after surgery. However, the measurement of vision is subjective and variable. Moreover, a patient's visual acuity is influenced by corneal aberrations, internal aberrations (due to cataracts) as well as retinal and neural factors.

With an aberrometer, one can specifically measure the aberrations of the (clouded) lens in the eye. This allows one to assess the effect of the cataract on visual acuity. Therefore, the investigators think the objective measurement of aberrations better reflects the optical distortions of cataract in the lens than visual acuity.

And although the indication for surgery is thus not optimal, the demand for excellent visual function is increasing among patients. In addition, the results and safety of this procedure have also continued to improve over the years. This may lower the indication for cataract surgery. However, both for the patient and in the context of value-driven care, it is important that a correct indication is made. This calls for a more objective indicator for cataract surgery.

The main aim of this project is to investigate whether an objective measurement of the optical quality of the eye can predict who is going to be satisfied with cataract surgery. The investigators do this by investigating the correlation of the objective measurement of the optical quality of the eye with the subjective change in visual functioning.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old,
* Diagnosis of cataract in both eyes,
* Based on informed consent, will undergo cataract surgery in both eyes (not necessarily immediately bilateral),
* Expected best-corrected visual acuity ≥ 0.7 in both eyes,
* Pupil diameter in mydriasis ≥4 mm and
* Implantation of a (standard) monofocal, toric monofocal or (non)toric Extended Depth of Focus artificial lens.

Exclusion Criteria:

* Insufficient understanding of the Dutch language to comply with study procedures,
* Spherical refraction of ≤-15 dioptres (due to impossibility of measurement with aberrometer),
* Corneal astigmatism of ≥3 dioptres (because of possible effect on reliability of straylight measurement),
* Implantation of a multifocal artificial lens (because the aberrometer [still] cannot properly determine the optical quality of this type of artificial lens),
* Cataract surgery of the second eye not performed 3 months after surgery of the first eye,
* Comorbidity (other than cataract) that may significantly affect vision or give prolonged duration of vision recovery, such as Fuchs' endothelial cell dystrophy, significant macular degeneration, glaucoma, diabetic maculo- or retinopathy, or an experienced cerebral vascular accident,
* A history of eye surgery (such as corneal refractive surgery and phakic lens implantation),
* An increased risk of complicated cataract surgery, such as lens (sub)luxation, brunescent cataract, posterior polar cataract and a history of trauma to the eye,
* Unable to be reliably measured with aberrometer or straylight meter, and
* A peroperative or postoperative complication that significantly affects vision and has not recovered within 3 months of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ophthalmic patients with cataracts in both eyes seeking surgery on them
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
log(VSX) | From enrollment to one year after cataract surgery
  preoperative aberrometry measurements, expressed as log(VSX)
log(s) | From enrollment to one year after cataract surgery
  preoperative straylight measurements, expressed as log(s)
preoperative Catquest-9SF score (expressed as Rasch score) | From enrollment to one year after cataract surgery
  preoperative Catquest-9SF score, expressed as Rasch score
postoperative Catquest-9SF score (expressed as Rasch score) | From enrollment to one year after cataract surgery
  postoperative Catquest-9SF score, expressed as Rasch score

CONTACTS AND LOCATIONS:
Overall Officials: Nic J Reus, MD, PhD, Principal Investigator — Amphia
Locations (1):
- Amphia, Breda, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No